CLINICAL TRIAL: NCT05479045
Title: A Combination Therapy Strategy to Prevent Anti-PD-1 Therapy Resistance in Metastatic Ovarian Cancer Patients
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: Coherus Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00005324
Record Dates: First submitted 2022-07-26; First posted 2022-07-29 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Ovarian Cancer Stage IV; Ovarian Cancer Stage III; Ovarian Cancer Stage 3
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NY-ESO-1 Peptide vaccine plus Toripalimab-tpzi (Experimental)
  Interventions: Biological: NY-ESO-1 Peptide vaccine; Drug: Toripalimab-tpzi

INTERVENTIONS:
Biological: NY-ESO-1 Peptide vaccine — 300 mcg of NY-ESO-1 peptide, 100 micrograms (mcg) granulocyte-macrophage colony-stimulating factor (GM-CSF) and 1 milliliter (mL) of Montanide ISA-51 adjuvant. The first two doses will be administered subcutaneously in a 2 week interval and thereafter, remaining three doses will be administered every 3 weeks.
Drug: Toripalimab-tpzi — 240 milligrams (mg), intravenously, every 3 weeks starting with the second dose of NY-ESO-1 Peptide vaccine
  Other Names: LOQTORZI

SUMMARY:
This is an open label, non-randomized, 2-stage phase II, single arm study to determine the efficacy of New York esophageal squamous cell carcinoma 1 (NY-ESO-1) peptide vaccine as a priming mechanism to prevent anti-PD1 resistance in patients with platinum-refractory stage III/IV ovarian cancer (OC).

ELIGIBILITY:
Inclusion Criteria:

1. Be able and willing to provide written and signed informed consent prior to performing any protocol-related procedures, including screening evaluations.
2. Women, 18 years or older, with stage III / IV platinum-refractory Ovarian Cancer (OC) (progressed on a platinum containing regimen within 6 months of therapy and adenocarcinoma histology) that can be evaluable by RECISTv1.1 criteria who progressed on standard treatment. Participants will be recruited irrespective of if they earlier received available FDA-approved therapies (including for participants with targetable mutations, such as BRCA mutations)
3. Subjects will be eligible for study entry based on the following diagnostic workup:

   1. History/physical examination within 28 days prior to registration.
   2. Imaging of target lesion(s) within 28 days prior to registration.
   3. Study-specific assessments:
   4. Recovery from effects of recent surgery, radiotherapy or chemotherapy.
   5. Free of active infection requiring antibiotics (with the exception of uncomplicated urinary tract infection).
   6. Any hormonal therapy directed at the malignant tumor must be discontinued at least one week prior to registration.
   7. Any other prior therapy directed at the malignant tumor including chemotherapy, targeted agents, biologic agents, immunologic agents, and any investigational agents, must be discontinued at least 4 weeks prior to registration (6 weeks for nitrosoureas or mitomycin C).
   8. Any prior radiation therapy must be completed at least 4 weeks prior to registration.
   9. At least 4 weeks must have elapsed since major surgery.
4. Subjects must have received and have progressed, are refractory, or are intolerant to standard platinum therapy. Subjects should not have received more than 2 prior lines of systemic therapy for recurrent or metastatic disease (including both standard of care and investigational therapies).
5. Subjects must have at least 1 lesion that is measurable using RECIST Version 1.1 guidelines.

   1. A previously irradiated lesion can be considered a target lesion if the lesion is well defined, measurable per RECIST Version 1.1, and has clearly progressed.
   2. Subjects undergoing fresh tumor biopsies must have additional non-target lesions that can be biopsied at acceptable risk as judged by the investigator (optional).
6. Subjects must consent to provide archived tumor specimens for correlative biomarker studies. Tumor tissue must be identified and availability confirmed prior to initiation of study therapy. In the setting where archival material is unavailable or unsuitable for use, subjects must consent and undergo fresh tumor biopsy.
7. All subjects are encouraged to consent to and provide both pretreatment and on-treatment (optional) tumor biopsies.
8. Eastern Cooperative Oncology Group (ECOG) Performance score of 2 or less.
9. In the opinion of the investigator likely to complete ≥ 8 weeks of treatment.
10. Adequate organ function as determined by:

    a) Hematological: i) Absolute neutrophil count (ANC) ≥ 1.0 × 109/L (1,000/mm3) ii) Absolute lymphocyte count (ALC) ≥ 0.5 × 109/L (500/mm3) iii) Platelet count ≥ 100 × 109/L (100,000/mm3) without transfusion support within first 2 weeks prior to first dose iv) Hemoglobin ≥ 9.0 g/dL without transfusion support within first 2 weeks prior to first dose b) Renal: i) Calculated creatinine clearance* (CrCl) or 24-hour urine CrCl > 50 mL/minute c) Hepatic: i) Total bilirubin ≤ 1.5 × upper limit of normal (ULN); for subjects with documented/suspected Gilbert's syndrome, bilirubin ≤ 3 × ULN ii) Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 × ULN (AST and/or ALT can be up to 5 × ULN in the presence of liver metastasis, but cannot be associated with concurrent elevated bilirubin)
11. Female subjects of childbearing potential who are sexually active with a nonsterilized male partner must use at least 1 highly effective method of contraception from screening, and must agree to continue using such precautions for 180 days after the final dose of investigational product. The male partner of the female subject must use male condom plus, if locally available, spermicide throughout this period. Cessation of contraception after this point should be discussed with a responsible physician. Not engaging in sexual activity for the duration of the study is an acceptable practice; however, periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of contraception.

    1. Females of childbearing potential are defined as those who are not surgically sterile (i.e., have not undergone bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy) or who are not postmenopausal (defined as 12 months with no menses without an alternative medical cause).
    2. A highly effective method of contraception is defined as one that results in a low failure rate (i.e., less than 1% per year) when used consistently and correctly.
    3. Subjects must refrain from breastfeeding while on study and for 180 days after the final dose of investigational product.

Exclusion Criteria:

1. Subjects who have received prior therapy with regimens containing nivolumab or CTLA-4, PD-L1, PD-L2 or PD-1 antagonists or any other antibody or drug specifically targeting T cell co-stimulation or immune checkpoint pathways.
2. Any condition that, in the opinion of the investigator, would interfere with evaluation of the investigational product or interpretation of subject safety or study results.
3. History of severe allergic reactions (i.e., Grade 4 allergy, anaphylactic reaction from which the subject did not recover within 6 hours of institution of supportive care) to any unknown allergens or any components of the study drug formulations.
4. Active or prior documented autoimmune disease (including inflammatory bowel disease, celiac disease, Wegener's granulomatosis) within the past 2 years. Subjects with childhood atopy or asthma, vitiligo, alopecia, Graves disease, Hashimoto disease, autoimmune diseases that will be consider stable by hormones /steroid replacement or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded.
5. Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or the follow-up period of an interventional study.
6. Receipt of any conventional or investigational anticancer therapy not otherwise specified above within 28 days prior to the first dose of the combination treatment; in the case of monoclonal antibodies, 28 days or 5 half-lives, whichever is shorter, prior to the first dose of the combination treatment.
7. Any concurrent chemotherapy, immunotherapy, or biologic or hormonal therapy for cancer treatment. Concurrent use of hormones for non-cancer-related conditions (e.g., insulin for diabetes and hormone replacement therapy) is acceptable.
8. Unresolved toxicities from prior anticancer therapy, defined as having not resolved to NCI CTCAE V5.0, Grade 0 or 1 with the exception of alopecia and laboratory values listed per the inclusion criteria. Subjects with irreversible toxicity that is not reasonably expected to be exacerbated by any of the investigational products may be included (e.g., hearing loss)
9. Current or prior use of immunosuppressive medication within 14 days prior to the first dose of any treatment regimen. The following are exceptions to this criterion:

   1. Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra-articular injection)
   2. Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or equivalent
   3. Steroids as premedication for hypersensitivity reactions (e.g., computerized tomography (CT) scan premedication)
10. History of primary immunodeficiency, solid organ transplantation, or tuberculosis.
11. Test results indicating active infection with hepatitis B or C defined by positive Hepatitis B DNA, Hepatitis C RNA or known HIV infection.
12. Receipt of live, attenuated vaccine within 28 days prior to the first dose of investigational products (NOTE: Subjects, if enrolled, should not receive live vaccine during the study and 180 days after the last dose of investigational products).
13. Pregnant or breastfeeding women.
14. Major surgery (as defined by the investigator) within 4 weeks prior to first dose of treatment regimen, or still recovering from prior surgery. Local surgery of isolated lesions for palliative intent is acceptable.
15. Other invasive malignancy within 2 years except for noninvasive malignancies such as cervical carcinoma in situ, non-melanomatous carcinoma of the skin, ductal carcinoma in situ of the breast or non invasive bladder carcinoma that has/have been surgically removed.
16. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, unstable angina pectoris, history of myocarditis, myocardial infarction ≤6 months, or congestive heart failure (as defined by New York Heart Association Functional Classification III or IV) requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring adverse events or compromise the ability of the subject to give written informed consent. In addition, participants with a left ventricular ejection fraction (LVEF) < 50% by echocardiogram will be excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Median Progression Free Survival | 2 years

SECONDARY OUTCOMES:
Median Overall Survival | 2 years
  per RECIST v1.1 and mRECIST v1.1
Overall Response Rate | 2 years
  based on irRECIST
Duration of Response | 2 years
  per RECIST v1.1 and mRECIST v1.1
Disease Control Rate | 2 years
  based on irRECIST
Incidence of Adverse Events (AE) | 2 years
  Safety and tolerability will be assessed by calculating the rates and frequencies of all AEs, serious adverse events (SAE), and any toxicities according to CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Samir N Khleif, MD, Principal Investigator — Georgetown University
Locations (2):
- United States (2):
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - John Theurer Cancer Center, Hackensack, New Jersey

IPD SHARING:
Plan to Share IPD: No